CLINICAL TRIAL: NCT00677469
Title: Low Doses of Cholestyramine in the Treatment of Hyperthyroidism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Golamhossein Ranjbar Omrani, Endocrine and Metabolism Research Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2590
Record Dates: First submitted 2008-05-12; First posted 2008-05-14 (Estimated); Last update posted 2008-05-14 (Estimated); Status verified 2008-05

CONDITIONS: Graves Disease
Keywords: Hyperthyroidism; Cholestyramine
MeSH Terms: conditions — Graves Disease; Hyperthyroidism | interventions — Cholestyramine Resin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- I (Experimental): Cholestyramine 2g BID, Methimazole 10mg TID, and Propranolol 20mg BID
  Interventions: Drug: Cholestyramine
- II (Experimental): Cholestyramine 1g BID, Methimazole 10mg TID, and Propranolol 20mg BID
  Interventions: Drug: Cholestyramine
- III (Placebo Comparator): Placebo powder 1g BID, Methimazole 10mg TID, and Propranolol 20mg BID
  Interventions: Drug: Placebo powder

INTERVENTIONS:
Drug: Cholestyramine — 2 grams BID
  Arms: I
Drug: Cholestyramine — 1 gram BID
  Arms: II
Drug: Placebo powder — 1 gram BID
  Arms: III

SUMMARY:
The enterohepatic circulation of thyroid hormones is increased in thyrotoxicosis.Bile-salt sequestrants (ionic exchange resins) bind thyroid hormones in the intestine and thereby increase their fecal excretion. Based on these observations, the use of cholestyramine has been tried. The present study evaluates the effect of low doses of cholestyramine as an adjunctive therapy in the management of hyperthyroidism

DETAILED DESCRIPTION:
The gastrointestinal tract has a role in thyroid physiology. Thyroid hormone is metabolized mainly in the liver, where it is conjugated to glucurunides and sulfates. These conjugation products are then excreted in the bile. Free hormones are released in the intestine and finally reabsorbed, completing the enterohepatic circulation of thyroid hormone. A very small portion of the daily production of thyroxin (T4) and triiodothyronine (T3), less than 10 percent, is excreted in the stool (1-3). In people with normal thyroid function, this pathway of T4 and T3 recirculation contributes so little to hormone availability that patients who have gastrointestinal disease or are receiving drugs that decrease T4 absorption do not have abnormal thyroid function (4). However, the thyrotoxic states are characterized by an increased enterohepatic circulation of thyroid hormones, as well as an increased urinary and fecal excretion of both conjugated and free T4 (5,6).

Cholestyramine, an ionic exchange resin sequesters T4 in the intestine and increases its fecal excretion. These phenomena were proven in hamsters in mid 1960s (7). Experimentally, it has been shown that 50 mg of cholestyramine can bind approximately 3000 μg of T4 (8) and therefore can enhance the clearance of thyroid hormones. Because of the increased enterohepatic circulation of thyroid hormones during hyperthyroidism, attempts have been made to sequester these hormones in the intestine using ionic exchange resins (9-13). Cholestyramine therapy has been studied in the treatment of thyrotoxicosis as an adjunctive therapy to thionamides, and has been found to decrease thyroid hormone levels rapidly. In several trials, cholestyramine in combination with methimazole (MMI) or propylthiouracil, caused a more rapid decline in thyroid hormone levels than standard therapy with thionamides alone (9-11,13). In all of these trials, cholestyramine was dosed at 4 grams orally two to four times a day.

This study was conducted to examine the efficacy of combination therapy of lower doses of cholestyramine with MMI and propranolol for treating patients with Graves' hyperthyroidism.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed hyperthyroid Graves' disease

Exclusion Criteria:

* If the patient had been treated previously
* diabetes, kidney, or liver disease

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2007-07; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Golamhossein Omrani, M.D., Study Chair — Endocrine and Metabolism Research Center
Locations (1):
- Endocrine and Metabolism Research Center, Shiraz, Fars, Iran

REFERENCES:
- [Derived] Kaykhaei MA, Shams M, Sadegholvad A, Dabbaghmanesh MH, Omrani GR. Low doses of cholestyramine in the treatment of hyperthyroidism. Endocrine. 2008 Aug-Dec;34(1-3):52-5. doi: 10.1007/s12020-008-9107-5. Epub 2008 Oct 23. PMID 18946743